CLINICAL TRIAL: NCT05060042
Title: Comparison of Whole Body Vibration With Bilateral Proprioceptive Training in Elderly Population
Brief Title: Comparison of Whole Body Vibration With Bilateral Proprioceptive Training in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Aneela Riaz
Record Dates: First submitted 2021-09-17; First posted 2021-09-28 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Elderly Population

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole body vibration group (Experimental): WBV will be provided with a frequency of 6-26Hz with amplitude of 1-3mm 4-5 bouts(60 sec each) for 3 times a week.
  Interventions: Other: Whole body vibration group
- Bilateral proprioceptive training Group (Active Comparator): Static balance training will be provided in first week for 3-4 times for 10 mints of single session. 3 times a week In 2nd and 3rd week dynamic balance training for 3 times with a session of 10 mints.
  In 4th week progressive balance training will be done with same frequency and duration.
  Tai chai exercises will be given for 20 mints 3 times a week
  Interventions: Other: Bilateral proprioceptive training

INTERVENTIONS:
Other: Whole body vibration group — WBV will be provided with a frequency of 6-26Hz with amplitude of 1-3mm 4-5 bouts(60 sec each) for 3 times a week
  Arms: Whole body vibration group
Other: Bilateral proprioceptive training — Static balance training will be provided in first week for 3-4 times for 10 mints of single session. 3 times a week In 2nd and 3rd week dynamic balance training for 3 times with a session of 10 mints.
  In 4th week progressive balance training will be done with same frequency and duration.
  Tai chai exercises will be given for 20 mints 3 times a week
  Arms: Bilateral proprioceptive training Group

SUMMARY:
The aim of this study is to conduct a randomized controlled trail to compare and analyze the effects of both whole body vibrator (WBV) and proprioceptive training through Tai Chi program on static and dynamic postural balance variables of the elderly population. The purpose of the study is to determine that whether whole body vibrator is more evident or proprioceptive training is more effective for promoting functional independency and improving balance in older adults. Hence distinguishing choices to prevent fall and advancing functional independency by using the appropriate intervention without using extreme loads.

DETAILED DESCRIPTION:
Elderly population is defined as 'people aged 65 or above'. Aging is a complex and challenging process of physiological changes and it is associated with decline of biological functions. Increasing age is linked with impairments in visual, proprioception, vestibular systems, decline in muscular strength and control of the lower limbs, balance/postural control, and of the mobility patterns which are known to be substantial hazards for fall, and these parameters have been found to be dynamically more disabled with getting older. Among all these factors, there is obvious decline in normal functioning and balance related issues, common in elderly population due to proprioceptive function loss that is the person is unable to sense his joint position and motion which ultimately results in mobility impairments.

Therefore, researchers have been looking for new approaches that are more feasible to improve the independence and physical mobility in older individuals and over the past decade the whole body vibrator (WBV) have been seeking attention for the beneficence of the elderly population. It is a neuromuscular training modality used to improve muscle strength, power, balance, mobility, cardiorespiratory rehabilitation, improves neuromuscular and musculoskeletal functions and general health both in healthy and as well as in orthopedic patients and neurologically diseased elderly population .Bilateral proprioceptive training is also used for impaired balance, proprioception loss and decreased ROM in elderly population. Proprioceptive receptors are present in our skin, muscles, tendons and joints with the help of which we can sense position and movement of limbs and trunk, sense of force and sense of heaviness in the absence of vision. The mechanoreceptors of the proprioception cause activation of central nervous system by initiating action potential through release of stored sodium in to the cells, this afferent sensory stimuli to the central nervous system is essential for the control of body movements

ELIGIBILITY:
Inclusion Criteria:

* Participants with balance and proprioception problems
* Those having BBS score between 21-54
* Intact cognition: MMSE >25

Exclusion Criteria:

* Subjects with recent trauma or any other neurodegenerative disorder.
* Subjects with cognitive and hearing impairments
* Subjects who cannot follow my command.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Time up and go test | Change from Baseline balance to 8th Weeks
  The assessment of functional mobility in community dwelling elderly population, is assessed precisely by a balance test called time up and go test.Time taken to complete the task is actually indicating the level of functional mobility. An elder participant taking less than 20 seconds to complete the task have been shown to be independent in ADLs. Time taken more than 30 seconds by an older subject, indicates more dependent in ADLs and requires assistive devices for ambulation.
Performance-Oriented Mobility Assessment (POMA): | Change from Baseline balance and gait to 8th Weeks
  • The Tinetti Performance Oriented Mobility Assessment (POMA) is a widely used clinical assessment tool that gives an insight into the abnormalities in balance and gait, and it has the ability to predict fall risk in elderly population.• This scale has a total maximum score of 28 in which there is 12 score of gait assessment and 16 score of balance assessment. The overall score of 25-28 indicates low fall risk, 19-24 represents moderate fall risk and <19 means there is high risk of fall in suspected elderly population. This scale has been declared has a valid and reliable tool to assess balance and gait impairments

CONTACTS AND LOCATIONS:
Overall Officials: Misbah ghous, MS, Principal Investigator — Riphah International University Islamabad
Locations (2):
- Pakistan (2):
  - Misbah Ghous, Rawalpindi, Islamabad
  - Pakistan General Railway Hospital, Rawalpindi, Islamabad

IPD SHARING:
Plan to Share IPD: No